CLINICAL TRIAL: NCT05266261
Title: Efficacy of Bisphosphonate Therapy on Postmenopausal Osteoporotic Women With and Without Diabetes: a Prospective Trial
Brief Title: Use of Ibandronate in Diabetic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yeouido St. Mary's Hospital (Other)
Collaborators: Samsung Medical Center (Other); Seoul National University Bundang Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SC18MEDV0024
Record Dates: First submitted 2022-02-20; First posted 2022-03-04 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-02

CONDITIONS: Osteoporosis, Postmenopausal; Type 2 Diabetes
MeSH Terms: conditions — Osteoporosis, Postmenopausal; Diabetes Mellitus, Type 2 | interventions — Ibandronic Acid; Calcium Carbonate; Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-diabetes (Active Comparator): postmenopausal women with normal glucose tolerance
  Interventions: Drug: Ibandronate Oral Tablet
- diabetes (Experimental): postmenopausal women with type 2 diabetes
  Interventions: Drug: Ibandronate Oral Tablet

INTERVENTIONS:
Drug: Ibandronate Oral Tablet — 150 mg of ibandronate + 24,000 IU of cholecalciferol
  Other Names: daily oral formulation of 1,250 mg of calcium carbonate + 1,000 IU of cholecalciferol

SUMMARY:
The purpose of this study is to examine whether monthly oral administration of ibandronate to postmenopausal osteoporosis patients with type 2 diabetes differs in safety and efficacy compared to patients without diabetes.

DETAILED DESCRIPTION:
There are two major considerations in the use of bisphosphonates in diabetic patients.

* The low rate of bone turnover in diabetic patients is at risk of side effects such as excessive inhibition of bone turnover associated with the use of bisphosphonates.
* A decrease in osteocalcin following bisphosphonate use may lead to deterioration of glucose metabolism.

The efficacy of ibandronate in T2DM is not thought to be significantly different based on previous studies, but there is few study on ibandronate.

ELIGIBILITY:
Inclusion Criteria:

* age of at least 55 years at the time of screening
* postmenopausal woman
* diagnosis of osteoporosis

Exclusion Criteria:

* history of osteoporosis treatment
* underlying disease (e.g., heart failure, liver disease, renal disease, or malignancy)
* the use of drugs that affect bone metabolism (e.g., steroids, immunosuppressants, gonadotropin-releasing hormone agonists, aromatase inhibitors, thiazolidinedione drugs, anticonvulsants, and antidepressants)
* history of adverse effects of bisphosphonate or difficulty taking the drug due to an inability to sit or the presence of upper gastrointestinal disease

Min Age: 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Bone mineral density | 1 year
  . Percentage change in dual-energy X-ray absorptiometry (DXA) bone mineral density (BMD) at the lumbar spine, total hip, and femoral neck, presented as least square mean and 95% confidence interval.

SECONDARY OUTCOMES:
Bone turnover markers | 6 month and 12 month
  Percentage change in bone turnover markers [Serum C-telopeptide (CTx) and procollagen type 1 N-terminal propeptide (P1NP) levels were measured by immunoassay methods using Elecsys kits - 07296355001V4 and 07296509001V4 (Roche Diagnostic Corp., Basel, Switzerland) ] presented as adjusted mean and 95% confidence interval using the generalized estimating equations for repeated measures analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Ki-Hyun Baek, M.D., Ph.D., Principal Investigator — Yeouido St. Mary's Hospital
Locations (1):
- Yeouido St.Mary's Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
The data that support the findings of this study are available from the corresponding author upon reasonable request.

REFERENCES:
- [Derived] Kim J, Kim KM, Lim S, Kang MI, Baek KH, Min YK. Efficacy of bisphosphonate therapy on postmenopausal osteoporotic women with and without diabetes: a prospective trial. BMC Endocr Disord. 2022 Apr 11;22(1):99. doi: 10.1186/s12902-022-01010-w. PMID 35410197